CLINICAL TRIAL: NCT06114004
Title: Phase I/II Randomized Clinical Trial of Selinexor Plus Gemcitabine in Selected Advanced Soft-tissue Sarcomas
Brief Title: Selinexor Plus Gemcitabine in Selected Advanced Soft-tissue Sarcoma (SeliSarc)
Acronym: SeliSarc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asociación Europea y Latinoamericana SELNET para la Investigación en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELNET-7-1
Record Dates: First submitted 2023-10-20; First posted 2023-11-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — selinexor; Gemcitabine

STUDY DESIGN:
Intervention Model Description: each cohort (1 and 2) receives the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gemcitabine + selinexor: (Experimental): Selinexor will be given at 60 mg once per week orally days 1, 8 and 15 every 21 days
  Gemcitabine will be given at the dose 1200 mg/m2 (10 mg/m2/min) days 1 and 8 every 21 days
  Interventions: Drug: Selinexor 20 MG; Drug: Gemcitabine

INTERVENTIONS:
Drug: Selinexor 20 MG — After having completed the Phase I part, the recommended dose for Phase II is 60mg Selinexor
  Other Names: KPT-330
Drug: Gemcitabine — Gemcitabine will be given at the dose 1200 mg/m2 (10 mg/m2/min) days 1 and 8 every 21 days.

SUMMARY:
Phase I-II, non-randomized, single-arm, open-label, multicenter, international clinical trial.

Patients with advanced soft-tissue sarcoma (leiomyosarcoma or malignant peripheral nerve sheath tumor) will receive selinexor in combination with gemcitabine.

DETAILED DESCRIPTION:
Phase I-II, non-randomized, single-arm, open-label, multicenter, international clinical trial.

Patients with advanced soft-tissue sarcoma (leiomyosarcoma or malignant peripheral nerve sheath tumor) will receive selinexor in combination with gemcitabine.

In the Phase I part safety and toxicity of the combination will be assessed using a 3+3 design. The recommended dose for the Phase II will be determined.

In the Phase II part there will be 2 different cohorts:

Cohort 1: Leiomyosarcoma (LMS) Cohort 2: Malignant peripheral nerve sheath tumor (MPNST)

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of any study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g. imaging tests), obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age: 18-80 years.
3. Histologic diagnosis of soft tissue sarcoma (leiomyosarcoma or malignant peripheral nerve sheath tumor) confirmed by central pathology review prior to enrolment with an archive tumor sample. A fresh paraffin embedded tumor tissue block must be provided for all subjects for biomarker analysis before and (when feasible) after treatment with investigational products.
4. Metastatic/advanced disease in progression in the last 6 months.
5. Patients have previously received at least one previous line of systemic therapy.
6. Measurable disease according to RECIST 1.1 criteria.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
8. Adequate hepatic, renal, cardiac, and hematologic function.
9. Laboratory tests as follows:

   * Absolute neutrophil count ≥ 1,500/mm³
   * Platelet count ≥ 100,000/mm³
   * Bilirubin ≤ 1.5 mg/dL
   * AST and ALT ≤ 2.5 times upper limit of normal
   * Creatinine ≤ 1.5 mg/dL 10. Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan.

11. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to enrollment and agree to use birth control measures during study treatment and for 3 months after its completion. Patients must not be pregnant or nursing at study entry. Women/men of reproductive potential must have agreed to use an effective contraceptive method.

Exclusion Criteria:

1. Three or more systemic treatment lines (including both chemotherapy and targeted therapy) for advanced disease (localized unresectable or metastatic).
2. Patients who have received any other anti-cancer therapy or investigational product in the last 21 days prior to enrollment.
3. Prior malignancy that required treatment or has shown evidence of recurrence (except for non-melanoma skin cancer, adequately treated cervical carcinoma in situ, superficial bladder carcinoma) during the 5 years prior to randomization. Cancer treated with curative intent for >5 years previously and without evidence of recurrence will be allowed.
4. Prior selinexor or another XPO1 inhibitor treatment.
5. Administration of a previous gemcitabine-containing treatment.
6. Any concurrent medical condition or disease (e.g. uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
7. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
8. Pregnant or breastfeeding females.
9. Body surface area (BSA) <1.4 m2 at baseline, calculated by the Du Bois(25) or Mosteller(26) method.
10. Life expectancy of less than 3 months.
11. Major surgery within 4 weeks prior to C1D1.
12. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or dysfunction that could interfere with absorption of study treatment.
13. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the NCCN CPGO for antiemesis and anorexia/cachexia (palliative care).
14. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent. 15. Presence of brain or central nervous system metastases, unless they are controlled (patients with treated and stable metastasis are eligible)
15. Presence of brain or central nervous system metastases, unless they are controlled (patients with treated and stable metastasis are eligible)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate (PFSR) | 6 months
  To evaluate the efficacy of the selinexor plus gemcitabine combination as measured by the progression-free survival rate (PFSR) at 6 months in patients with selected advanced soft-tissue sarcomas.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  Overall survival (OS): OS is defined as the time between the date of first dose and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.
Overall response rate (ORR) according to RECIST 1.1 | 6 months
  Overall Response Rate (ORR): ORR is defined as the number of subjects with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) divided by the number of response evaluable subjects.
Evaluate the efficacy according to Choi response | 6 months
  Efficacy measured through tumor response according to Choi criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow-up until tumor progression.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 6 months
  Safety profile of the experimental treatment, through assessment of adverse event type, incidence, severity, time of appearance, related causes, as well as physical explorations and laboratory tests. Toxicity will be graded and tabulated by using CTCAE 5.0.
Patients's quality of life (QoL) | 6 months
  Quality of life will be measured with European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire 30

CONTACTS AND LOCATIONS:
Overall Officials: Javier MD Martín Broto, Study Director — Hospital Universitario Fundación Jiménez Díaz
Locations (11):
- Spain (11):
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clinico Universitario Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner JG, Sullivan DM. CRM1-mediated nuclear export of proteins and drug resistance in cancer. Curr Med Chem. 2008;15(26):2648-55. doi: 10.2174/092986708786242859. PMID 18991627
- [Background] Das A, Wei G, Parikh K, Liu D. Selective inhibitors of nuclear export (SINE) in hematological malignancies. Exp Hematol Oncol. 2015 Mar 1;4:7. doi: 10.1186/s40164-015-0002-5. eCollection 2015. PMID 25745591
- [Background] Yao Y, Dong Y, Lin F, Zhao H, Shen Z, Chen P, Sun YJ, Tang LN, Zheng SE. The expression of CRM1 is associated with prognosis in human osteosarcoma. Oncol Rep. 2009 Jan;21(1):229-35. PMID 19082467
- [Background] Gravina GL, Senapedis W, McCauley D, Baloglu E, Shacham S, Festuccia C. Nucleo-cytoplasmic transport as a therapeutic target of cancer. J Hematol Oncol. 2014 Dec 5;7:85. doi: 10.1186/s13045-014-0085-1. PMID 25476752
- [Background] Abdul Razak AR, Mau-Soerensen M, Gabrail NY, Gerecitano JF, Shields AF, Unger TJ, Saint-Martin JR, Carlson R, Landesman Y, McCauley D, Rashal T, Lassen U, Kim R, Stayner LA, Mirza MR, Kauffman M, Shacham S, Mahipal A. First-in-Class, First-in-Human Phase I Study of Selinexor, a Selective Inhibitor of Nuclear Export, in Patients With Advanced Solid Tumors. J Clin Oncol. 2016 Dec;34(34):4142-4150. doi: 10.1200/JCO.2015.65.3949. Epub 2016 Oct 31. PMID 26926685
- [Background] Gounder MM, Zer A, Tap WD, Salah S, Dickson MA, Gupta AA, Keohan ML, Loong HH, D'Angelo SP, Baker S, Condy M, Nyquist-Schultz K, Tanner L, Erinjeri JP, Jasmine FH, Friedlander S, Carlson R, Unger TJ, Saint-Martin JR, Rashal T, Ellis J, Kauffman M, Shacham S, Schwartz GK, Abdul Razak AR. Phase IB Study of Selinexor, a First-in-Class Inhibitor of Nuclear Export, in Patients With Advanced Refractory Bone or Soft Tissue Sarcoma. J Clin Oncol. 2016 Sep 10;34(26):3166-74. doi: 10.1200/JCO.2016.67.6346. Epub 2016 Jul 25. PMID 27458288
- [Background] Gounder MM, Razak AA, Somaiah N, Chawla S, Martin-Broto J, Grignani G, Schuetze SM, Vincenzi B, Wagner AJ, Chmielowski B, Jones RL, Riedel RF, Stacchiotti S, Loggers ET, Ganjoo KN, Le Cesne A, Italiano A, Garcia Del Muro X, Burgess M, Piperno-Neumann S, Ryan C, Mulcahy MF, Forscher C, Penel N, Okuno S, Elias A, Hartner L, Philip T, Alcindor T, Kasper B, Reichardt P, Lapeire L, Blay JY, Chevreau C, Valverde Morales CM, Schwartz GK, Chen JL, Deshpande H, Davis EJ, Nicholas G, Groschel S, Hatcher H, Duffaud F, Herraez AC, Beveridge RD, Badalamenti G, Eriksson M, Meyer C, von Mehren M, Van Tine BA, Gotze K, Mazzeo F, Yakobson A, Zick A, Lee A, Gonzalez AE, Napolitano A, Dickson MA, Michel D, Meng C, Li L, Liu J, Ben-Shahar O, Van Domelen DR, Walker CJ, Chang H, Landesman Y, Shah JJ, Shacham S, Kauffman MG, Attia S. Selinexor in Advanced, Metastatic Dedifferentiated Liposarcoma: A Multinational, Randomized, Double-Blind, Placebo-Controlled Trial. J Clin Oncol. 2022 Aug 1;40(22):2479-2490. doi: 10.1200/JCO.21.01829. Epub 2022 Apr 8. PMID 35394800
- [Background] Ishizawa J, Kojima K, Hail N Jr, Tabe Y, Andreeff M. Expression, function, and targeting of the nuclear exporter chromosome region maintenance 1 (CRM1) protein. Pharmacol Ther. 2015 Sep;153:25-35. doi: 10.1016/j.pharmthera.2015.06.001. Epub 2015 Jun 3. PMID 26048327
- [Background] De Cesare M, Cominetti D, Doldi V, Lopergolo A, Deraco M, Gandellini P, Friedlander S, Landesman Y, Kauffman MG, Shacham S, Pennati M, Zaffaroni N. Anti-tumor activity of selective inhibitors of XPO1/CRM1-mediated nuclear export in diffuse malignant peritoneal mesothelioma: the role of survivin. Oncotarget. 2015 May 30;6(15):13119-32. doi: 10.18632/oncotarget.3761. PMID 25948791
- [Background] Nakayama R, Zhang YX, Czaplinski JT, Anatone AJ, Sicinska ET, Fletcher JA, Demetri GD, Wagner AJ. Preclinical activity of selinexor, an inhibitor of XPO1, in sarcoma. Oncotarget. 2016 Mar 29;7(13):16581-92. doi: 10.18632/oncotarget.7667. PMID 26918731
- [Background] Moysan E, Bastiat G, Benoit JP. Gemcitabine versus Modified Gemcitabine: a review of several promising chemical modifications. Mol Pharm. 2013 Feb 4;10(2):430-44. doi: 10.1021/mp300370t. Epub 2012 Oct 8. PMID 22978251
- [Background] Plunkett W, Huang P, Gandhi V. Preclinical characteristics of gemcitabine. Anticancer Drugs. 1995 Dec;6 Suppl 6:7-13. doi: 10.1097/00001813-199512006-00002. PMID 8718419
- [Background] Siena L, Pace E, Ferraro M, Di Sano C, Melis M, Profita M, Spatafora M, Gjomarkaj M. Gemcitabine sensitizes lung cancer cells to Fas/FasL system-mediated killing. Immunology. 2014 Feb;141(2):242-55. doi: 10.1111/imm.12190. PMID 24128051
- [Background] Garcia-Del-Muro X, Lopez-Pousa A, Maurel J, Martin J, Martinez-Trufero J, Casado A, Gomez-Espana A, Fra J, Cruz J, Poveda A, Meana A, Pericay C, Cubedo R, Rubio J, De Juan A, Lainez N, Carrasco JA, de Andres R, Buesa JM; Spanish Group for Research on Sarcomas. Randomized phase II study comparing gemcitabine plus dacarbazine versus dacarbazine alone in patients with previously treated soft tissue sarcoma: a Spanish Group for Research on Sarcomas study. J Clin Oncol. 2011 Jun 20;29(18):2528-33. doi: 10.1200/JCO.2010.33.6107. Epub 2011 May 23. PMID 21606430
- [Background] Sonnenblick A, Eleyan F, Peretz T, Ospovat I, Merimsky O, Sella T, Peylan-Ramu N, Katz D. Gemcitabine in combination with paclitaxel for advanced soft-tissue sarcomas. Mol Clin Oncol. 2015 Jul;3(4):829-832. doi: 10.3892/mco.2015.545. Epub 2015 Apr 16. PMID 26171190
- [Background] Kashyap T, Argueta C, Unger T, Klebanov B, Debler S, Senapedis W, Crochiere ML, Lee MS, Kauffman M, Shacham S, Landesman Y. Selinexor reduces the expression of DNA damage repair proteins and sensitizes cancer cells to DNA damaging agents. Oncotarget. 2018 Jul 20;9(56):30773-30786. doi: 10.18632/oncotarget.25637. eCollection 2018 Jul 20. PMID 30112106
- [Background] Kazim S, Malafa MP, Coppola D, Husain K, Zibadi S, Kashyap T, Crochiere M, Landesman Y, Rashal T, Sullivan DM, Mahipal A. Selective Nuclear Export Inhibitor KPT-330 Enhances the Antitumor Activity of Gemcitabine in Human Pancreatic Cancer. Mol Cancer Ther. 2015 Jul;14(7):1570-81. doi: 10.1158/1535-7163.MCT-15-0104. Epub 2015 May 1. PMID 25934708
- [Background] Park KS, Han BG, Lee KH, Kim DS, Kim JM, Jeon H, Kim HS, Suh SW, Lee EH, Kim SY, Lee BI. Depletion of nucleophosmin via transglutaminase 2 cross-linking increases drug resistance in cancer cells. Cancer Lett. 2009 Feb 18;274(2):201-7. doi: 10.1016/j.canlet.2008.09.007. Epub 2008 Oct 11. PMID 18851895
- [Background] Hill R, Rabb M, Madureira PA, Clements D, Gujar SA, Waisman DM, Giacomantonio CA, Lee PW. Gemcitabine-mediated tumour regression and p53-dependent gene expression: implications for colon and pancreatic cancer therapy. Cell Death Dis. 2013 Sep 5;4(9):e791. doi: 10.1038/cddis.2013.307. PMID 24008735
- [Background] Gravina GL, Tortoreto M, Mancini A, Addis A, Di Cesare E, Lenzi A, Landesman Y, McCauley D, Kauffman M, Shacham S, Zaffaroni N, Festuccia C. XPO1/CRM1-selective inhibitors of nuclear export (SINE) reduce tumor spreading and improve overall survival in preclinical models of prostate cancer (PCa). J Hematol Oncol. 2014 Oct 5;7:46. doi: 10.1186/1756-8722-7-46. PMID 25284315
- [Background] Gordon N, Kleinerman ES. The role of Fas/FasL in the metastatic potential of osteosarcoma and targeting this pathway for the treatment of osteosarcoma lung metastases. Cancer Treat Res. 2009;152:497-508. doi: 10.1007/978-1-4419-0284-9_29. PMID 20213411
- [Background] Martin-Broto J, Pousa AL, de Las Penas R, Garcia Del Muro X, Gutierrez A, Martinez-Trufero J, Cruz J, Alvarez R, Cubedo R, Redondo A, Maurel J, Carrasco JA, Lopez-Martin JA, Sala A, Meana JA, Ramos R, Martinez-Serra J, Lopez-Guerrero JA, Sevilla I, Balana C, Vaz A, De Juan A, Alemany R, Poveda A. Randomized Phase II Study of Trabectedin and Doxorubicin Compared With Doxorubicin Alone as First-Line Treatment in Patients With Advanced Soft Tissue Sarcomas: A Spanish Group for Research on Sarcoma Study. J Clin Oncol. 2016 Jul 1;34(19):2294-302. doi: 10.1200/JCO.2015.65.3329. Epub 2016 May 16. PMID 27185843
- [Background] Maki RG, Wathen JK, Patel SR, Priebat DA, Okuno SH, Samuels B, Fanucchi M, Harmon DC, Schuetze SM, Reinke D, Thall PF, Benjamin RS, Baker LH, Hensley ML. Randomized phase II study of gemcitabine and docetaxel compared with gemcitabine alone in patients with metastatic soft tissue sarcomas: results of sarcoma alliance for research through collaboration study 002 [corrected]. J Clin Oncol. 2007 Jul 1;25(19):2755-63. doi: 10.1200/JCO.2006.10.4117. PMID 17602081
- [Background] Seddon B, Strauss SJ, Whelan J, Leahy M, Woll PJ, Cowie F, Rothermundt C, Wood Z, Benson C, Ali N, Marples M, Veal GJ, Jamieson D, Kuver K, Tirabosco R, Forsyth S, Nash S, Dehbi HM, Beare S. Gemcitabine and docetaxel versus doxorubicin as first-line treatment in previously untreated advanced unresectable or metastatic soft-tissue sarcomas (GeDDiS): a randomised controlled phase 3 trial. Lancet Oncol. 2017 Oct;18(10):1397-1410. doi: 10.1016/S1470-2045(17)30622-8. Epub 2017 Sep 4. PMID 28882536
- [Background] Du Bois D, Du Bois EF. A formula to estimate the approximate surface area if height and weight be known. 1916. Nutrition. 1989 Sep-Oct;5(5):303-11; discussion 312-3. No abstract available. PMID 2520314
- [Background] Mosteller RD. Simplified calculation of body-surface area. N Engl J Med. 1987 Oct 22;317(17):1098. doi: 10.1056/NEJM198710223171717. No abstract available. PMID 3657876
- [Background] Seddon B, Scurr M, Jones RL, Wood Z, Propert-Lewis C, Fisher C, Flanagan A, Sunkersing J, A'Hern R, Whelan J, Judson I. A phase II trial to assess the activity of gemcitabine and docetaxel as first line chemotherapy treatment in patients with unresectable leiomyosarcoma. Clin Sarcoma Res. 2015 May 16;5:13. doi: 10.1186/s13569-015-0029-8. eCollection 2015. PMID 25987978
- [Background] Ordonez JL, Martins AS, Osuna D, Madoz-Gurpide J, de Alava E. Targeting sarcomas: therapeutic targets and their rational. Semin Diagn Pathol. 2008 Nov;25(4):304-16. doi: 10.1053/j.semdp.2008.07.005. PMID 19013896
- [Background] Gilbert JA, Salavaggione OE, Ji Y, Pelleymounter LL, Eckloff BW, Wieben ED, Ames MM, Weinshilboum RM. Gemcitabine pharmacogenomics: cytidine deaminase and deoxycytidylate deaminase gene resequencing and functional genomics. Clin Cancer Res. 2006 Mar 15;12(6):1794-803. doi: 10.1158/1078-0432.CCR-05-1969. PMID 16551864
- [Background] Khan MA, Srivastava SK, Bhardwaj A, Singh S, Arora S, Zubair H, Carter JE, Singh AP. Gemcitabine triggers angiogenesis-promoting molecular signals in pancreatic cancer cells: Therapeutic implications. Oncotarget. 2015 Nov 17;6(36):39140-50. doi: 10.18632/oncotarget.3784. PMID 25970774
- [Background] Kondo S, Ueno H, Hashimoto J, Morizane C, Koizumi F, Okusaka T, Tamura K. Circulating endothelial cells and other angiogenesis factors in pancreatic carcinoma patients receiving gemcitabine chemotherapy. BMC Cancer. 2012 Jun 25;12:268. doi: 10.1186/1471-2407-12-268. PMID 22731825
- [Background] Martin-Broto J, Redondo A, Valverde C, Vaz MA, Mora J, Garcia Del Muro X, Gutierrez A, Tous C, Carnero A, Marcilla D, Carranza A, Sancho P, Martinez-Trufero J, Diaz-Beveridge R, Cruz J, Encinas V, Taron M, Moura DS, Luna P, Hindi N, Lopez-Pousa A. Gemcitabine plus sirolimus for relapsed and progressing osteosarcoma patients after standard chemotherapy: a multicenter, single-arm phase II trial of Spanish Group for Research on Sarcoma (GEIS). Ann Oncol. 2017 Dec 1;28(12):2994-2999. doi: 10.1093/annonc/mdx536. PMID 29045512
- [Background] Kamran SC, Howard SA, Shinagare AB, Krajewski KM, Jagannathan JP, Hornick JL, Ramaiya NH. Malignant peripheral nerve sheath tumors: prognostic impact of rhabdomyoblastic differentiation (malignant triton tumors), neurofibromatosis 1 status and location. Eur J Surg Oncol. 2013 Jan;39(1):46-52. doi: 10.1016/j.ejso.2012.09.001. Epub 2012 Oct 18. PMID 23084090
- [Background] Le Guellec S, Macagno N, Velasco V, Lamant L, Lae M, Filleron T, Malissen N, Cassagnau E, Terrier P, Chevreau C, Ranchere-Vince D, Coindre JM. Loss of H3K27 trimethylation is not suitable for distinguishing malignant peripheral nerve sheath tumor from melanoma: a study of 387 cases including mimicking lesions. Mod Pathol. 2017 Dec;30(12):1677-1687. doi: 10.1038/modpathol.2017.91. Epub 2017 Jul 28. PMID 28752843
- [Background] Luzar B, Shanesmith R, Ramakrishnan R, Fisher C, Calonje E. Cutaneous epithelioid malignant peripheral nerve sheath tumour: a clinicopathological analysis of 11 cases. Histopathology. 2016 Jan;68(2):286-96. doi: 10.1111/his.12756. Epub 2015 Jul 28. PMID 26096054
- [Background] Kolberg M, Holand M, Agesen TH, Brekke HR, Liestol K, Hall KS, Mertens F, Picci P, Smeland S, Lothe RA. Survival meta-analyses for >1800 malignant peripheral nerve sheath tumor patients with and without neurofibromatosis type 1. Neuro Oncol. 2013 Feb;15(2):135-47. doi: 10.1093/neuonc/nos287. Epub 2012 Nov 15. PMID 23161774
- [Background] Hirbe AC, Dahiya S, Miller CA, Li T, Fulton RS, Zhang X, McDonald S, DeSchryver K, Duncavage EJ, Walrath J, Reilly KM, Abel HJ, Pekmezci M, Perry A, Ley TJ, Gutmann DH. Whole Exome Sequencing Reveals the Order of Genetic Changes during Malignant Transformation and Metastasis in a Single Patient with NF1-plexiform Neurofibroma. Clin Cancer Res. 2015 Sep 15;21(18):4201-11. doi: 10.1158/1078-0432.CCR-14-3049. Epub 2015 Apr 29. PMID 25925892
- [Background] Zhang M, Wang Y, Jones S, Sausen M, McMahon K, Sharma R, Wang Q, Belzberg AJ, Chaichana K, Gallia GL, Gokaslan ZL, Riggins GJ, Wolinksy JP, Wood LD, Montgomery EA, Hruban RH, Kinzler KW, Papadopoulos N, Vogelstein B, Bettegowda C. Somatic mutations of SUZ12 in malignant peripheral nerve sheath tumors. Nat Genet. 2014 Nov;46(11):1170-2. doi: 10.1038/ng.3116. Epub 2014 Oct 12. PMID 25305755
- [Background] Lee W, Teckie S, Wiesner T, Ran L, Prieto Granada CN, Lin M, Zhu S, Cao Z, Liang Y, Sboner A, Tap WD, Fletcher JA, Huberman KH, Qin LX, Viale A, Singer S, Zheng D, Berger MF, Chen Y, Antonescu CR, Chi P. PRC2 is recurrently inactivated through EED or SUZ12 loss in malignant peripheral nerve sheath tumors. Nat Genet. 2014 Nov;46(11):1227-32. doi: 10.1038/ng.3095. Epub 2014 Sep 21. PMID 25240281
- [Background] De Raedt T, Beert E, Pasmant E, Luscan A, Brems H, Ortonne N, Helin K, Hornick JL, Mautner V, Kehrer-Sawatzki H, Clapp W, Bradner J, Vidaud M, Upadhyaya M, Legius E, Cichowski K. PRC2 loss amplifies Ras-driven transcription and confers sensitivity to BRD4-based therapies. Nature. 2014 Oct 9;514(7521):247-51. doi: 10.1038/nature13561. Epub 2014 Aug 13. PMID 25119042
- [Background] Al-Ezzi E, Gounder M, Watson G, Mazzocca A, D'Angelo SP, Bravetti J, Wang H, Abdul Razak A, Vincenzi B. Selinexor, a First in Class, Nuclear Export Inhibitor for the Treatment of Advanced Malignant Peripheral Nerve Sheath Tumor. Oncologist. 2021 Apr;26(4):e710-e714. doi: 10.1002/onco.13692. Epub 2021 Feb 17. PMID 33512749
- [Background] Kolberg M, Bruun J, Murumagi A, Mpindi JP, Bergsland CH, Holand M, Eilertsen IA, Danielsen SA, Kallioniemi O, Lothe RA. Drug sensitivity and resistance testing identifies PLK1 inhibitors and gemcitabine as potent drugs for malignant peripheral nerve sheath tumors. Mol Oncol. 2017 Sep;11(9):1156-1171. doi: 10.1002/1878-0261.12086. Epub 2017 Jul 5. PMID 28556483
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] van der Graaf WT, Blay JY, Chawla SP, Kim DW, Bui-Nguyen B, Casali PG, Schoffski P, Aglietta M, Staddon AP, Beppu Y, Le Cesne A, Gelderblom H, Judson IR, Araki N, Ouali M, Marreaud S, Hodge R, Dewji MR, Coens C, Demetri GD, Fletcher CD, Dei Tos AP, Hohenberger P; EORTC Soft Tissue and Bone Sarcoma Group; PALETTE study group. Pazopanib for metastatic soft-tissue sarcoma (PALETTE): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2012 May 19;379(9829):1879-86. doi: 10.1016/S0140-6736(12)60651-5. Epub 2012 May 16. PMID 22595799
- [Background] Wang Z, Shi N, Naing A, Janku F, Subbiah V, Araujo DM, Patel SR, Ludwig JA, Ramondetta LM, Levenback CF, Ramirez PT, Piha-Paul SA, Hong D, Karp DD, Tsimberidou AM, Meric-Bernstam F, Fu S. Survival of patients with metastatic leiomyosarcoma: the MD Anderson Clinical Center for targeted therapy experience. Cancer Med. 2016 Dec;5(12):3437-3444. doi: 10.1002/cam4.956. Epub 2016 Nov 23. PMID 27882721
- [Background] Kantidakis G, Litiere S, Neven A, Vinches M, Judson I, Schoffski P, Wardelmann E, Stacchiotti S, D'Ambrosio L, Marreaud S, van der Graaf WTA, Kasper B, Fiocco M, Gelderblom H. Efficacy thresholds for clinical trials with advanced or metastatic leiomyosarcoma patients: A European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group meta-analysis based on a literature review for soft-tissue sarcomas. Eur J Cancer. 2021 Sep;154:253-268. doi: 10.1016/j.ejca.2021.06.025. Epub 2021 Jul 20. PMID 34298376
- [Background] Van Glabbeke M, Verweij J, Judson I, Nielsen OS; EORTC Soft Tissue and Bone Sarcoma Group. Progression-free rate as the principal end-point for phase II trials in soft-tissue sarcomas. Eur J Cancer. 2002 Mar;38(4):543-9. doi: 10.1016/s0959-8049(01)00398-7. PMID 11872347
- [Background] Sobczuk P, Teterycz P, Czarnecka AM, Switaj T, Kosela-Paterczyk H, Kozak K, Falkowski S, Rutkowski P. Systemic Treatment for Advanced and Metastatic Malignant Peripheral Nerve Sheath Tumors-A Sarcoma Reference Center Experience. J Clin Med. 2020 Sep 29;9(10):3157. doi: 10.3390/jcm9103157. PMID 33003503

DOCUMENTS (1):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT06114004/Prot_000.pdf